CLINICAL TRIAL: NCT04647760
Title: Packaging and Disseminating the JOIN for ME Program in Low-Income Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: Brown University (Other); University of North Carolina, Chapel Hill (Other); Tufts University (Other); Brandeis University (Other)
Responsible Party: Principal Investigator, Elissa Jelalian, Professor; Associate Director, Weight Control & Diabetes Research Center, The Miriam Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5U18DP006429-02 (NIH)
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Obesity
Keywords: Pediatric; Pediatric obesity; Pediatric overweight; Community-based; Behavioral weight loss
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Hybrid-implementation effectiveness design incorporating a delayed-treatment design for treatment group assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Other): Participants will start the intervention immediately upon study enrollment.
  Interventions: Behavioral: JOIN for ME
- Delayed treatment (Other): Participants will start the intervention 4-months post enrollment.
  Interventions: Behavioral: JOIN for ME

INTERVENTIONS:
Behavioral: JOIN for ME — JOIN for ME is an empirically tested, effective weight management program for children ages 6-12 years.The curriculum includes 16 weekly in person sessions followed by 4 biweekly and 4 monthly maintenance sessions for a 10-month program. Weekly meetings are attended by the parent/caregiver and child, and occur at a location within their community setting (public housing or patient-centered medical home). Each session is 60 minutes and led by a certified Community Health Worker, with a private weigh-in for each dyad prior to the start of each session. Key behavioral targets include self-monitoring of dietary intake and physical activity, limiting LESS foods, limiting screen time, and weekly attendance. A family-based incentive structure is incorporated into the program such that parents/caregivers reinforce their children for achieving goals. Due to the COVID-19 pandemic, in-person sessions will be conducted virtually until it is safe to resume in-person group sessions.

SUMMARY:
One in five children in the United States have obesity, and under-served populations are differentially impacted by both obesity and its related health consequences. Thus, community-based programs that improve the dissemination of effective obesity treatments are needed within low income settings. The current study aims to test the effectiveness of an evidence-based, community centered program, JOIN for ME, in two types of community settings: housing authorities and patient-centered medical homes. Children between the ages of 6-12 years old and who meet study eligibility criteria will be enrolled in the study and participate in the JOIN for ME weight control intervention. Participants will be assigned to active or delayed treatment conditions (4-month delay) but all participants will receive the JOIN for ME program. The program will be delivered in English or Spanish. Primary outcomes include change in child and parent weight status and health-related quality of life.

DETAILED DESCRIPTION:
The U.S. Preventive Services Task Force (USPSTF) recently reissued a Grade B recommendation, initially made in 2010, for clinicians to screen children ages 6-18 years for obesity and refer identified youth to comprehensive, multi-component programs with >26 contact hours that include nutrition and physical activity targets and are supported by behavioral strategies. Re-issue of this recommendation highlights the continued importance of comprehensive family-based obesity treatment programs with broad accessibility. The challenge in meeting this objective is the lack of community-based obesity treatments for children. The majority of children in the U.S. do not receive evidence-based treatment of obesity, with few such programs available to youth from low-income backgrounds.

There are multiple efforts underway to broaden both the empirical support for, and accessibility of, pediatric weight management interventions. One such strategy is implementation within the primary care setting as families are already accustomed to attending visits for medical concerns and because physicians are important drivers of health behavior change. An alternative strategy, also with high impact potential, is embedding interventions in established organizations within the communities in which families live, thereby decreasing logistical barriers (e.g. transportation) and enhancing program credibility.

The JOIN for ME program, developed as a collaboration between United HealthGroup and Y-USA, is an empirically tested, effective pediatric weight control intervention for children ages 6-12 years that is delivered by facilitators within a community setting and potentially scalable nationally. The primary aim of this study is to test the effectiveness of the the JOIN for ME intervention in two different types of community setting, housing authorities and patient-centered medical homes, with the intention to increase equity and access to care for families in low-income settings. To accomplish this aim, formative qualitative work was conducted during 2019-2020 with key community stakeholders and families within the targeted community settings. The formative work resulted in adapting "participant facing" intervention materials and tools as well as the development of systems to connect families with local community resources. These developments will be implemented in intervention delivery as a means of increasing acceptability of the intervention and assessing its potential for broader scale dissemination within community settings. Further, certified Community Health Workers (CHWs) will deliver the proposed intervention given their ability to serve as intermediaries between healthcare systems and the community.

A total of 128 children (ages 6-12) with BMI > 85th% will be enrolled in this study and receive the JOIN for ME weight control intervention. The intervention will be delivered in English or Spanish. Participants will be assigned to active or delayed treatment conditions (4-month delay) based on an a priori set of rules pertaining to recruitment strategies and timeline. Evaluation of primary outcomes, change in child and parent weight status and health-related quality of life (HRQL), will be obtained at baseline, 4 months, and 10 months.

The following hypotheses will be tested:

1. Children who receive the JOIN for ME program immediately will demonstrate greater decreases in percent over median BMI and zBMI from baseline to 4 months compared to those in the delayed treatment onset prior to receiving the intervention.
2. Children who receive the JOIN for ME program immediately will demonstrate improvements in HRQL from baseline to 4 months compared to those in the delayed treatment onset.

ELIGIBILITY:
Inclusion Criteria:

* be 6 to 12 years old
* have a BMI > 85th percentile
* have at least one caregiver available to provide consent and participate in sessions
* speak English or Spanish
* agree to study participation and delayed treatment onset if applicable.

Exclusion Criteria:

* either the child or the parent is currently involved in another weight loss program
* have a medical condition that would interfere with the prescribed dietary plan or participation in physical activity
* are developmentally delayed such that the intervention materials will not be appropriate
* are in treatment for or diagnosed with a major psychiatric disorder, including an eating disorder

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 111 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Patient Outcome - Change in child weight status | Baseline, post-intensive treatment 1 (4 months), post-maintenance treatment 2 (10 months)
  Change in Body Mass Index (BMI, kg/m2)-for age-percentile
Patient Outcome - Change in parent weight status | Baseline, post-intensive treatment 1 (4 months), post-maintenance treatment 2 (10 months)
  Change in Body Mass Index (BMI, kg/m2)
Patient Outcome - Change in child health-related quality of life (HRQL) | Baseline, post-intensive treatment 1 (4 months), post-maintenance treatment 2 (10 months)
  Obesity-specific child self-report measure, Size Me Up
Patient Outcome - Change in parent health-related quality of life (HRQL) | Baseline, post-intensive treatment 1 (4 months), post-maintenance treatment 2 (10 months)
  Obesity-specific parent self-report measure, Sizing Them Up

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Jelalian, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- Weight Management and Diabetes Research Center, The Miriam Hospital/Alpert Medical School of Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified data set will be submitted to a data repository or to an investigator created website, if a central repository is not available. IPD which underlie results in a publication will be included in the repository.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be submitted to a repository or otherwise made available within 12 months of completion of the grant or coincident with publication of a manuscript based on the study findings, whichever is sooner. Long-term preservation will be described once a repository/website for deidentified data has been identified and the details are known.
Access Criteria: Access criteria will be provided once a repository/wesbite for deidentified data has been identified and the details are known.

REFERENCES:
- [Derived] Darling KE, Hayes JF, Evans EW, Seifer R, Elwy AR, Jelalian E. Implementation of the JOIN for ME Program for Families from Low-Income Backgrounds: The Use of Theory-Driven Formative Evaluation: Rhode Island CORD 3.0. Child Obes. 2021 Sep;17(S1):S22-S29. doi: 10.1089/chi.2021.0172. PMID 34569847
- [Derived] Jelalian E, Evans W, Darling KE, Seifer R, Vivier P, Goldberg J, Wright C, Tanskey L, Warnick J, Hayes J, Shepard D, Tuttle H, Elwy AR. Protocol for the Rhode Island CORD 3.0 Study: Adapting, Testing, and Packaging the JOIN for ME Family-Based Childhood Obesity Program in Low-Income Communities. Child Obes. 2021 Sep;17(S1):S11-S21. doi: 10.1089/chi.2021.0179. PMID 34569839

DOCUMENTS (1):
  • Informed Consent Form (2021-04-02): https://cdn.clinicaltrials.gov/large-docs/60/NCT04647760/ICF_000.pdf